CLINICAL TRIAL: NCT02475590
Title: Laparoscopic Sleeve Gastrectomy Versus Roux-en-Y Gastric Bypass for Morbidly Obese Patients: a Prospective Randomized Clinical Trial
Brief Title: Laparoscopic Sleeve Gastrectomy Versus Roux-en-Y Gastric Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IHU Strasbourg (Other)
Collaborators: IRCAD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-A01590-55
Record Dates: First submitted 2015-05-26; First posted 2015-06-18 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Morbid Obesity
Keywords: Sleeve gastrectomy; Roux-en-Y gastric bypass; Excess weight loss; Quality of life
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleeve gastrectomy (Experimental): Laparoscopic sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Roux-en-Y gastric bypass (Experimental): Laparoscopic Roux-en-Y gastric bypass
  Interventions: Procedure: Laparoscopic Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy
  Arms: Sleeve gastrectomy
Procedure: Laparoscopic Roux-en-Y gastric bypass — Laparoscopic Roux-en-Y gastric bypass
  Arms: Roux-en-Y gastric bypass

SUMMARY:
Prospective randomized clinical trial aiming to compare laparoscopic Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG) with primary outcome on excess weight loss, and secondary outcomes on nutritional status, glycolipid profile, quality of life and pain assessments.

DETAILED DESCRIPTION:
No consensus is proposed by the Medical and Surgical societies to define and / or prioritize surgical procedures in obesity surgery. Indications are based on patient's age, sex, dietary habits, the importance of overweight and associated comorbidities and even if rarely admitted, based on knowledge of surgical teams and the cost of interventions. Given the decrease of gastric banding procedures, Roux-en-Y gastro-jejunal bypass is often considered the reference procedure.

The gastric bypass, developed in the 60s, is performed laparoscopically since the early 90s. It allows for a 60% to 70% excess weight loss with control over 75% of comorbidities. It is recommended to follow these patients long-term because late complications can occur. These patients require ongoing information and regular monitoring. They must also have a hyper-protein diet and a vitamin substitute long-term (multivitamins, vitamin B12, calcium ...).

The Sleeve gastrectomy (SG) arises as an alternative to RYGB. It was classically proposed to patients with a BMI greater than 60 and significant comorbidities since the procedure let to a significant weight reduction in patients for whom any other procedure was too difficult to perform. The quality of the weight loss achieved in these patients has led many teams to analyze the results of this intervention without conducting an additional procedure. It appears from the literature that even performed alone, SG presents many benefits.

To clarify the role of sleeve gastrectomy in the bariatric procedures range, the investigators propose to conduct a prospective randomized study to compare laparoscopic sleeve gastrectomy to Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 and < 60 kg/m2
* No contraindication to any of the procedures
* No contraindication to general anesthesia
* No known addiction
* Patient able to provide informed consent

Exclusion Criteria:

* Contraindication to general anesthesia
* Known psychiatric pathology
* Pregnancy
* Previous major digestive surgery
* Immunosuppressive treatment including corticoids
* Coagulopathy (INR>1.5) or platelets < 50 000/µl
* Anemia (Hb<10g/dl)
* Severe comorbidity
* Malabsorptive disease or gastro-intestinal disease
* Myocardial infarction in previous year, angina, cardiac failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss at 3 years | At 36 months
  % of excess weight loss
Change in excess weight loss | At 1, 3, 6, 12, months and every year for 10 years
  % of excess weight loss

SECONDARY OUTCOMES:
Nutritional status and vitamin deficiency | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Albumin
Nutritional status and vitamin deficiency | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Pre-albumin
Nutritional status and vitamin deficiency | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Vitamin A
Nutritional status and vitamin deficiency | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Vitamin D
Nutritional status and vitamin deficiency | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Vitamin B9
Nutritional status and vitamin deficiency | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Vitamin B12
Glycolipid profile | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Fasting plasma glucose
Glycolipid profile | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Serum insulin
Glycolipid profile | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  HbA1c
Glycolipid profile | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Triglycerides
Glycolipid profile | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Cholesterol (total, HDL, LDL)
Quality of life (Moorehead-Ardelt II, Gastro-intestinal Quality of Life Index (GIQLI)) | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Moorehead-Ardelt II, Gastro-intestinal Quality of Life Index (GIQLI)
Pain (visual analog scale) | At 1, 3, 6, 12, 18, 24, 30 and 36 months
  Pain assessment (visual analog scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Marescaux, MD, Principal Investigator — Strasbourg university hospital, IRCAD, IHU Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, Strasbourg, France

REFERENCES:
- [Background] Vix M, Liu KH, Diana M, D'Urso A, Mutter D, Marescaux J. Impact of Roux-en-Y gastric bypass versus sleeve gastrectomy on vitamin D metabolism: short-term results from a prospective randomized clinical trial. Surg Endosc. 2014 Mar;28(3):821-6. doi: 10.1007/s00464-013-3276-x. Epub 2013 Nov 7. PMID 24196556
- [Background] Vix M, Diana M, Liu KH, D'Urso A, Mutter D, Wu HS, Marescaux J. Evolution of glycolipid profile after sleeve gastrectomy vs. Roux-en-Y gastric bypass: results of a prospective randomized clinical trial. Obes Surg. 2013 May;23(5):613-21. doi: 10.1007/s11695-012-0827-5. PMID 23207829
- [Derived] Ignat M, Vix M, Imad I, D'Urso A, Perretta S, Marescaux J, Mutter D. Randomized trial of Roux-en-Y gastric bypass versus sleeve gastrectomy in achieving excess weight loss. Br J Surg. 2017 Feb;104(3):248-256. doi: 10.1002/bjs.10400. Epub 2016 Nov 30. PMID 27901287